CLINICAL TRIAL: NCT06878664
Title: Randomized Interval Assessment Trial of Lu177-Dotatate Every 8 Versus Every 16 Weeks in Slowly Progressive G1-2 Advanced Midgut Neuroendocrine Tumors (NETs) to Lower TOxicity
Brief Title: Randomized Interval Assessment Trial of Lu177-Dotatate in Slowly Progressive G1-2 Advanced Midgut Neuroendocrine Tumors
Acronym: RIALTO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: Grupo Español de Tumores Neuroendocrinos y Endocrinos (GETNE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RLTTio2023 / GETNE T2421; 2024-517921-14-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-04; First posted 2025-03-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Grade1-2 Advanced Midgut Neuroendocrine Tumors (NETs)
Keywords: midgut; Neuroendocrine Tumors; Lu177-Dotatate
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate; Lutetium; Lutetium-177; copper dotatate CU-64; amino-acid, glucose, and electrolyte solution; lanreotide

STUDY DESIGN:
Intervention Model Description: RIALTO is an a randomized, prospective, international, open-label, phase III - I trial comparing a less intensive RLT regimen (4 cycles of 177Lu-Dotatate (7·4 GBq/cycle) every 16 weeks) versus the conventional one (4 cycles of 177Lu-Dotatate (7·4 GBq/cycle) every 8 weeks).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 177Lu-Dotatate every 16 weeks (Experimental): Experimental arm:
  1. Treatment with 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 16 weeks (q16w) x 4 cycles
  2. Renal protection starting 30 minutes before targeted radioligand therapy (RLT) lasting 4 hours (iv amino acid solution of 14.4-20g of lysine and 14.9-20.7g of arginine in 1 to 2 liters of solution)
  3. Long-acting standard doses of SSA (Lanreotide autogel 120 mg subcutaneous or Octreotide LAR 30 mg intramuscular, starting 24h after RLT every 4 weeks during RLT (q16w interval SSA administration should be adjusted to RLT administrations so that SSA is always given 24h after each RLT dose and at least 4 weeks prior to next RLT administration cycle) and q4w following last RLT administration until disease progression.
  Interventions: Drug: 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 16 weeks (q8w) x 4 cycles; 2) and 3) as in the experimental arm.; Drug: Amino acid solution; Drug: Lanreotide (Autogel formulation) or Octreotide LAR
- 177Lu-Dotatate every 8 weeks (Active Comparator): 1. Treatment with 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 8 weeks (q8w) x 4 cycles
  2. Renal protection starting 30 minutes before targeted radioligand therapy (RLT) lasting 4 hours (iv amino acid solution of 14.4-20g of lysine and 14.9-20.7g of arginine in 1 to 2 liters of solution);
  3. Long-acting standard doses of SSA (Lanreotide autogel 120 mg subcutaneous or Octreotide LAR 30 mg intramuscular, starting 24h after RLT every 4 weeks during RLT (q8w interval SSA administration should be adjusted to RLT administrations so that SSA is always given 24h after each RLT dose and at least 4 weeks prior to next RLT administration cycle) and q4w following last RLT administration until disease progression
  Interventions: Drug: 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 8 weeks (q8w) x 4 cycles; 2) and 3) as in the experimental arm.; Drug: Amino acid solution; Drug: Lanreotide (Autogel formulation) or Octreotide LAR

INTERVENTIONS:
Drug: 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 16 weeks (q8w) x 4 cycles; 2) and 3) as in the experimental arm. — Treatment with 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 16 weeks
  177Lu-Dotatate, a radiopharmaceutical medicine which is an somatostatin analogue derived from octreotide that complexes via DOTA with non-carrier added (n.c.a) 177Lu radioconjugate.
  177Lu-Dotatate will be supplied as a 370 MBq/mL solution for infusion. One mL of solution contains 370 MBq The total amount of radioactivity per single-dose vial is 7 400 MBq at the date and time of infusion. Given the fixed volumetric activity of 370 MBq/mL at the date and time of calibration, the volume of the solution in the vial ranges between 20.5 and 25.0 mL in order to provide the required amount of radioactivity at the date and time of infusion of lutetium (177Lu) oxodotreotide at the date and time of calibration.
  Other Names: 177Lu-DOTA0-Tyr 3-Octreotate, 177Lu-DOTATE; LUTATHERA, lutetium (177Lu) oxodotreotide
  Arms: 177Lu-Dotatate every 16 weeks
Drug: 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 8 weeks (q8w) x 4 cycles; 2) and 3) as in the experimental arm. — Treatment with 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 8 weeks (q8w) x 4 cycles 177Lu-Dotatate, a radiopharmaceutical medicine which is an somatostatin analogue derived from octreotide that complexes via DOTA with non-carrier added (n.c.a) 177Lu radioconjugate.
  Synonyms are:
  177Lu-DOTA0-Tyr 3-Octreotate, 177Lu-DOTATE LUTATHERA, lutetium (177Lu) oxodotreotide 177Lu-Dotatate will be supplied as a 370 MBq/mL solution for infusion One mL of solution contains 370 MBq The total amount of radioactivity per single-dose vial is 7 400 MBq at the date and time of infusion. Given the fixed volumetric activity of 370 MBq/mL at the date and time of calibration, the volume of the solution in the vial ranges between 20.5 and 25.0 mL in order to provide the required amount of radioactivity at the date and time of infusion of lutetium (177Lu) oxodotreotide at the date and time of calibration.
  Arms: 177Lu-Dotatate every 8 weeks
Drug: Amino acid solution — Renal protection starting 30 minutes before RLT and lasting 4 hours (iv) amino acid solution of 14.4-20 g of lysine and 14.9-20.7 g of arginine in 1 to 2 liters of solution)
Drug: Lanreotide (Autogel formulation) or Octreotide LAR — Long-acting standard doses of SSA (Lanreotide autogel 120 mg subcutaneous (sc) or Octreotide LAR 30 mg im, starting 24h after RLT and every 4 weeks during RLT (q16w interval SSA administration should be adjusted to RLT administrations so that SSA is always given 24h after each RLT dose and at least 4 weeks prior to next RLT administration cycle) and q4w following last RLT administration until disease progression.

SUMMARY:
This is a randomized Phase II/late phase I de-escalation clinical trial with approved investigational medicinal products in new use condition, low intervention.

Disease under study Patients with unresectable or metastatic, slowly progressive, well-differentiated (Grade1 and Grade2), somatostatin receptor-positive midgut neuroendocrine tumors (GEP-NETs).

It is planned to randomize 166 patients with a histologically confirmed diagnosis of slowly progressive grade 1 or grade 2 advanced midgut neuroendocrine tumors (NETs) candidates to receive 177Lu-Dotatate targeted radioligand therapy (RLT). Patients are required to have SSTR+ disease, as evidenced on somatostatin receptor imaging. Patients will be randomized into two arms:

1. control arm: regimen 177Lu-Dotatate every 8 weeks (q8w)
2. experimental arm: regimen 177Lu-Dotatate every 16 weeks (q16w)

Research hypothesis: Less intensive somatostatin-receptor (SST) targeted radioligand therapy (RLT) (7.4 GBq/cycle 177Lu-Dotatate every 16 weeks x 4 cycles) is associated with less severe hematological toxicities and may mitigate the risk to develop therapy-related myeloid neoplasms (t-MN) with similar antitumor efficacy in slowly growing gastrointestinal grade 1-2 NETs.

DETAILED DESCRIPTION:
1. Rationale The main hypothesis is less intensive somatostatin-receptor (SST) targeted radioligand therapy (RLT) (7.4 GBq/cycle 177Lu-Dotatate every 16 weeks x 4 cycles) is associated with less severe hematological toxicities and may mitigate the risk to develop therapy-related myeloid neoplasms (t-MN) with similar antitumor efficacy in slowly growing gastrointestinal grade 1-2 NETs.
2. Objectives Primary Objectives

   -To demonstrate decreased serious hematological toxicity with a less intensive RLT regimen in slowly progressive advanced Grade 1-2 midgut NETs.

   Secondary Objectives
   * To show comparable efficacy (clinical, hormonal and radiological response, progression-free survival and overall survival) of the less intensive RLT regimen (cycles q16w) versus the conventional one (cycles q8w). To compare the rate of clonal hematopoiesis among study arms (baseline and post-treatment) and assess its potential value to predict the risk of therapy-related myeloid neoplasms (t-MN).
   * To compare the duration of ≥ Grade 2 hematological toxicity (median and percentage rate of > 6 month duration)
   * To show decreased overall toxicity of the less intensive RLT regimen (cycles q16w) versus the conventional one (cycles q8w) Exploratory Objectives
   * To explore other predictive factors for toxicity and efficacy
   * To explore the tolerance of the subsequent systemic line of treatment Pattern of progression and modality of diagnosis
3. Main Trial Endpoints The primary endpoint for the RIALTO trial is the rate of Grade 2-5 hematological toxicity (worst per patient) from initiation of treatment with RLT up to 24 months thereafter according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5)
4. Secondary Trial Endpoints

   * Best hormonal response
   * Best radiological response
   * Duration of response (DoR)
   * Objective response rate (ORR)
   * Disease control rate (DCR)
   * Progression-free survival (PFS) (investigator assessed)
   * Overall survival (date of randomization to death from any cause)
   * Worst grade non-hematological toxicity per patient
   * Rate of clonal hematopoiesis by Next-Generation Sequencing (NGS) of ctDNA
   * Number of RLT cycles and cumulative dose received
   * Treatment compliance analyzing treatment delays and interruptions due to toxicity, rate of patients completing planned schedule, time from first to last RLT dose
   * Rate of Grade 2-5 hematological toxicity (worst per patient) from initiation of treatment with RLT up to 3, 6 or 12 months after the last PRRT
   * PFS will also be centrally assessed based only on morphological imaging (CT/MRI scans), regardless of SRI-PET scan results.
   * PFS will also be centrally assessed based on both morphological (CT/MRI scans) and functional imaging.
   * PFS will also be assessed based only on morphological imaging (CT/MRI scans), functional imaging and clinically progression of the functional syndrome, defined as unequivocal worsening of the functioning syndrome at the investigator criteria Secondary Safety endpoints
   * Adverse events (AE) and serious adverse events (SAE).
   * Treatment-related AEs (TRAEs).
   * Patients reported outcomes through the EORTC QLQ-C30 and GINET21 questionnaires.
   * Rate of myeloid neoplasms
   * Incidence of severe infection/sepsis (antibiotics prescription, hospitalization)
   * Duration of adverse events ≥ Grade 2
   * Rate of adverse events ≥ Grade 2 under subsequent next line of systemic treatment Exploratory endpoints
   * Correlation between clinical factors, radiomics and molecular determinants and toxicity/efficacy of 177Lu-Dotatate using mathematical models including artificial intelligence algorithms.
   * Tolerance of the subsequent systemic line of treatment
   * Pattern of progression (mesenteric, peritoneum, bone vs others) and modality of diagnosis
5. Trial Design RIALTO is an a randomized, prospective, international, open-label, phase III - I trial comparing a less intensive RLT regimen 4 cycles of 177Lu-Dotatate (7·4 GBq/cycle) every 16 weeks) versus the conventional one (4 cycles of 177Lu-Dotatate (7·4 GBq/cycle) every 8 weeks)
6. Trial Population It is planned to randomize 166 patients with a histologically confirmed diagnosis of slowly progressive grade 1 or grade 2 advanced midgut neuroendocrine tumors (NETs) candidates to receive 177Lu-Dotatate targeted radioligand therapy (RLT). Patients are required to have SSTR+ disease, as evidenced on somatostatin receptor imaging. Patients with a large SRI+ mesenteric mass with abdominal-dominant disease judged by the investigator to be a midgut NET will also be eligible. Patients will be randomized into two arms: control (regimen 177Lu-Dotatate every 8 weeks) and experimental (regimen 177Lu-Dotatate every 16 weeks).
7. Study Treatments

Patients will be randomized in a 1:1 ratio to experimental or control arms respectively:

Experimental arm:

1. Treatment with 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 16 weeks (q16w) x 4 cycles
2. Renal protection starting 30 minutes before targeted radioligand therapy (RLT) lasting 4 hours (iv amino acid solution of 14.4-20g of lysine and 14.9-20.7g of arginine in 1 to 2 liters of solution)
3. Long-acting standard doses of SSA (Lanreotide autogel 120 mg subcutaneous or Octreotide LAR 30 mg intramuscular, starting 24h after RLT every 4 weeks during RLT (q16w interval SSA administration should be adjusted to RLT administrations so that SSA is always given 24h after each RLT dose and at least 4 weeks prior to next RLT administration cycle) and q4w following last RLT administration until disease progression.

Control arm:

1. Treatment with 177Lu-Dotatate (7.4 Gigabecquerel/cycle) during 30 min intravenous infusion every 8 weeks (q8w) x 4 cycles
2. Renal protection starting 30 minutes before targeted radioligand therapy (RLT) lasting 4 hours (iv amino acid solution of 14.4-20g of lysine and 14.9-20.7g of arginine in 1 to 2 liters of solution);
3. Long-acting standard doses of SSA (Lanreotide autogel 120 mg subcutaneous or Octreotide LAR 30 mg intramuscular, starting 24h after RLT every 4 weeks during RLT (q8w interval SSA administration should be adjusted to RLT administrations so that SSA is always given 24h after each RLT dose and at least 4 weeks prior to next RLT administration cycle) and q4w following last RLT administration until disease progression

8. Ethical Considerations

The study will be conducted in accordance with the principles of the Helsinki Declaration Adopted by the 18th World Medical Assembly, Helsinki, Finland, June 1964 updated to its latest version Fortaleza, Brazil, October 2013. With the Good Clinical Practice (GCP) standards issued by the Working Party on Medicinal Product Efficacy of the European Economic Community (1990) (CPMP / ICH / 135/95).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have histologically confirmed diagnosis of unresectable, advanced or metastatic midgut NETs (originated in the jejunum-ileum or right colon) who are candidates to receive 177Lu-Dotatate targeted radioligand therapy (RLT) and SSA. Patients with a large SRI+ mesenteric mass with abdominal-dominant disease judged by the investigator to be a midgut NET will also be eligible.
2. Ki-67 index ≤ 20%.
3. Disease progression per RECIST v1.1 within 36 months prior to study entry,
4. Patients may be treatment naïve (first-line) or have received prior systemic therapy except for any type of prior RLT (not restricted to 177Lu-Dotatate).
5. In somatostatin receptor (SSTR) imaging all RECIST v1.1 evaluable target lesions and non-target lesions need to be SSTR positive (SSTR+) as defined by equal or above the liver uptake (this includes lesions of at least 10 mm in diameter in CT or MRI). If an FDG PET is performed (not mandatory), all FDG PET positive lesions should also be somatostatin receptor positive in SSRT imaging (see guidance Appendix 10).
6. Measurable disease according to RECIST v1.1 criteria (Appendix 3)
7. Adequate organ function (hematological, renal and liver) based upon meeting all of the following laboratory criteria:

   * Neutrophil count (ANC) ≥ 2.000/mm3
   * Platelet count ≥ 75 × 109/L
   * Hemoglobin ≥ 8 g/dL
   * Serum bilirubin ≤ 3.0 × upper limit of normal (ULN) or ≤ 3 × ULN for subjects with Gilbert's disease
   * Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
   * Creatinine clearance (CrCl) ≥ 50 mL/min as estimated by the Cockroft-Gault formula or as measured by 24-hour urine collection (GFR can also be used instead of CrCl). Note: renal tract obstruction is not allowed.
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 xULN for subjects with liver metastases
8. Karnofsky performance status (KPS) scale ≥ 70%
9. Patient information and signing of the consent form, Institutional Review Board(IRB)/Independent Ethics Committee (IEC) approved, before any study-specific procedure. The patient must be able and willing to cooperate in monitoring study visits and procedures.
10. Patients ≥ 18 years of age.
11. Recovery to Grade ≤ 1 from any adverse event (AE) from prior treatment (excluding alopecia and/or asthenia).
12. Life expectancy ≥ 12 months.
13. Patients with health coverage (public or private), that includes coverage for patients enrolled in clinical trials, to both study treatments and determinations/procedures.
14. Female subject must provide a negative urine pregnancy test at screening, and must agree to use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%; refer to Appendix 4) for the duration of the study treatment and for 7 months after the final dose of study treatment. Sexually active men must agree to use the male condom during the study and until at least 7 months after the last administration of treatment. Additionally, it is recommended that your female partner of childbearing age use a highly effective method of contraception.
15. Subject agrees not to participate in another interventional study while on treatment in the present study.

Exclusion Criteria:

1. Patients who have known hypersensitivity to lutetium-177 (177Lu), oxodotreotide, DOTA, somatostatin analogues, lysine, arginine, or any excipient/derivative of these agents
2. Prior external beam radiation therapy (EBRT) to more than 25% of the bone marrow
3. Prior whole liver internal radiation therapy (SIRT)
4. Prior radioligand therapy (RLT) (not restricted to 177Lu-Dotatate).
5. Prior major surgery, systemic therapy, embolization or other locoregional treatments within 4 weeks of study entry
6. Patients who have a known active Hepatitis B (e.g., HBsAg reactive) or active hepatitis C (e.g., HCV RNA [qualitative] is detected). Patients who have a known active history of human immunodeficiency virus (HIV) infection (HIV 1 or 2).
7. Other known malignancies unless cured or definitively treated with no evidence of recurrence for 3 years
8. Serious non-malignant disease (e.g. psychiatric, infectious, autoimmune, cardiovascular or dementia), that may interfere with the objectives of the trial or with the safety or compliance of the patient, as judged by the investigator.
9. Female patients must agree not to breastfeed or donate ovules starting at screening and throughout the study period, and for at least 7 months after the final study drug administration.
10. Male patients must agree not to donate sperm starting at screening and throughout the study period, and for at least 4 months after the final study drug administration.
11. Pregnancy or lactation. Men and women should not procreate during study treatment and until seven months after the final study drug administration.
12. For female patients of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male patients who are not surgically sterile and have female partners of childbearing potential that do not agree to use a medically accepted and highly effective birth control method (i.e. those with a failure rate less than 1%; refer to Appendix 4) for the duration of the study treatment and for 7 months after the final dose of study treatment
13. Patient under guardianship or curatorship or deprived of liberty by a judicial or administrative decision or patient unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Grade 2-5 hematological toxicity | Throughout the study period, from initiation of treatment with RLT up to 24 months
  The primary endpoint for the RIALTO trial is the frequency of Grade 2-5 hematological toxicity (worst per patient) from initiation of treatment with RLT up to 24 months thereafter according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5)

SECONDARY OUTCOMES:
Best hormonal response | 24 months
  Best hormonal response defined as greatest decrease, or >30% decrease, of chromogranin A and 5HIAA from baseline if baseline levels were >2x ULN or 5xULN
Best radiological response | 24 months
  Best radiological response according to local investigator RECIST V1.1
Duration of response (DoR) | Throughout the study period, from initiation of treatment with RLT up to 24 months
  Duration of response (DoR) according to local investigator RECIST v1.1. Time from first response (CR or PR), according to ORR definition for the trial, to the date of the documented PD as determined using RECIST v1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment.
Objective response rate (ORR) | Throughout the study period, from initiation of treatment with RLT up to 24 months
  Objective response rate (ORR) according to local investigator RECIST v1.1. Assessed by the investigator through imaging follow-up (CT scan/MRI) using RECIST v1.1 (Appendix 3). This will be considered as the percentage/proportion of randomized patients with complete response (CR) or partial response (PR) as their overall best response throughout the study period. The investigator will report the change in size of tumors as compared with baseline, before the first dose of study treatment.
Disease control rate (DCR) | Throughout the study period, from initiation of treatment with RLT up to 24 months
  Disease control rate (DCR) RECIST v1.1 according to local investigator RECIST v1.1. Assessed by the investigator through imaging follow-up (CT scan/MRI) using RECIST v1.1. This will be considered as the percentage/proportion of randomized patients with complete response (CR) or partial response (PR) as their overall best response throughout the study period. The investigator will report the change in size of tumors as compared with baseline, before the first dose of study treatment.
Progression-free survival (PFS) | Throughout the study period, up to 3 months from radomization
  Progression-free survival (PFS) (investigator assessed) defined as the time between randomization date and disease progression according to RECIST v1.1 or death from any cause (primary analysis of PFS) .PFS will be censored at the date of the last adequate tumor assessment if no PFS event is observed prior to the analysis cut-off date.
Progression-free survival (PFS) | Throughout the study period, up to 12 months from radomization
  Progression-free survival (PFS) (investigator assessed) defined as the time between randomization date and disease progression according to RECIST v1.1 or death from any cause (primary analysis of PFS). PFS will be censored at the date of the last adequate tumor assessment if no PFS event is observed prior to the analysis cut-off date.
Progression-free survival (PFS) | Throughout the study period, up to 24 months from radomization
  Progression-free survival (PFS) (investigator assessed) defined as the time between randomization date and disease progression according to RECIST v1.1 or death from any cause (primary analysis of PFS) .PFS will be censored at the date of the last adequate tumor assessment if no PFS event is observed prior to the analysis cut-off date.
Overall survival | Throughout the study period, up to 6 months from radomization
  Overall survival defined as the time elapsed from randomization until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Overall survival | Throughout the study period, up to 12 months from radomization
  Overall survival defined as the time elapsed from randomization until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Overall survival | Throughout the study period, up to 18 months from radomization
  Overall survival defined as the time elapsed from randomization until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Overall survival | Throughout the study period, up to 24 months from radomitation
  Overall survival defined as the time elapsed from randomization until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact.
Worst grade non-hematological toxicity per patient | Throughout the study period, up to 24 months
  Percentage of patients with Non-hematological toxicity. Non-hematological toxicity: defined as worst grade non-hematological toxicity per patient according to NCI-CTCAE v 5.0 criteria.
Rate of clonal hematopoiesis | Throughout the study period, at baseline
  Rate of clonal hematopoiesis by Next-Generation Sequencing (NGS) of ctDNA calculated by mutations frequency in ctDNA samples
Rate of clonal hematopoiesis | Throughout the study period, up to 3 months from the start of treatment of the study
  Rate of clonal hematopoiesis by Next-Generation Sequencing (NGS) of ctDNA calculated by mutations frequency in ctDNA
Rate of clonal hematopoiesis | Throughout the study period, up to 12 months from the start of treatment of the study
  Rate of clonal hematopoiesis by Next-Generation Sequencing (NGS) of ctDNA calculated by mutations frequency in ctDNA samples
Rate of clonal hematopoiesis | Throughout the study period, up to 24 months from the start of treatment of the study
  Rate of clonal hematopoiesis by Next-Generation Sequencing (NGS) of ctDNA calculated by mutations frequency in ctDNA samples.
Number of RLT cycles per patient | Throughout the study period, up to 24 month
  Number of RLT cycles per patient
Acumulative dose received each patient | Throughout the study period up to 24 month
  Number acumulative dose received each patient
Treatment compliance analyzing treatment delays and interruptions due to toxicity | Throughout the study period, time from first to last RLT dose
  Treatment compliance analyzing treatment delays and interruptions due to toxicity, rate of patients completing planned schedule, time from first to last RLT dose
Rate of Grade 2-5 hematological toxicity (worst per patient) | Throughout the study period, from initiation of treatment with RLT up to12 months after the last PRRT
  Rate of Grade 2-5 hematological toxicity (worst per patient) from initiation of treatment with RLT up to 12 months after the last PRRT
PFS centralized based only on morphological imaging | Throughout the study period, up to 24 mounth from radomization
  PFS will also be centrally assessed according to RECIST 1.1 based only on morphological imaging (CT/MRI scans), regardless of SRI-PET scan results.
PFS will also be centralized on both morphological and functional imaging. | Throughout the study period up to 24 mounth from radomization
  Progression-free survival will also be centrally assessed according to RECIST 1.1 based on both morphological (CT/MRI scans) and functional imaging.
PFS will also be assessed according to RECIST 1.1 based only on morphological imaging, functional imaging and clinically progression of the functional syndrome | Throughout the study period, up to 24 mounth from radomization
  PFS will also be assessed according to RECIST 1.1 based only on morphological imaging (CT/MRI scans), functional imaging and clinically progression of the functional syndrome, defined as unequivocal worsening of the functioning syndrome at the investigator criteria
Adverse events (AE) and serious adverse events (SAE). | Throughout the study period. 24 months
  Number patients that suffered a Adverse event (AE) or serious adverse events (SAE) specific
Treatment-related AEs (TRAEs). | Throughout the study period, 24 month
  Number Treatment-related AEs (TRAEs).
Patients reported outcomes through the EORTC QLQ-C30 and GINET21 questionnaires. | Throughout the study period, 24 months
  Patients reported outcomes through the EORTC QLQ-C30 and GINET21 questionnaires.
Rate of myeloid neoplasms | Throughout the study period
  Porcentatge patients with myeloid neoplasms
Incidence of severe infection/sepsis | Throughout the study period
  Incidence of severe infection/sepsis (antibiotics prescription, hospitalization)
Rate of adverse events ≥ Grade 2 | Throughout the study period
  Rate of adverse events ≥ Grade 2 under subsequent next line of systemic treatment
Duration of adverse events ≥ Grade 2 | Throughout the study period
  Duration of adverse events ≥ Grade 2 (median, %>6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Garcia Carbonero Garcia Carbonero, M.D., Ph.D., Study Director — Hospital Universitario 12 de Octubre; Eric Baudin Baudin, M.D., Ph.D., Study Director — Gustave Roussy, Cancer Campus, Grand Paris
Locations (21):
- France (8):
  - Centre François BACLESSE, Caen, Caen
  - Chu Dijon, Dijon, Dijon
  - Hospital Center University De Lille, Lille, Lille
  - Hospices civiles de Lyon, Lyon, Lyon
  - Institut Paoli Calmette, Marseille, Marseille
  - Hopital BEAUJON, Clichy, Paris
  - Hopital COCHIN, Paris, Paris
  - Centre Eugène MARQUIS, Rennes, Rennes
- Spain (13):
  - Hospital Universitario de Burgos, Burgos, Balearic Islands
  - Hospital Universitari Vall d'Hebrón, Barcelona, Barcelona
  - Instituto Catalán de Oncología - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Virgen de las Nieves de Granada, Granada, Granada
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No